CLINICAL TRIAL: NCT07222007
Title: Association of Induction Agent Choice With Early Mortality and Prognostic Outcomes in Critically Ill Patients: A Large-Scale Retrospective Cohort Analysis
Brief Title: Induction Agent Choice With Early Mortality and Prognostic Outcomes in Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Zeliha Alicikus (Other Government)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor-Investigator, Zeliha Alicikus, Assoc. prof. dr, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: Tolga-01
Record Dates: First submitted 2025-10-21; First posted 2025-10-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Critically Ill; Intubation Complication; Oxygenation; Airway Management; Propofol; Ketamine
Keywords: intubation, critically ill patients, airway management
MeSH Terms: conditions — Critical Illness | interventions — Intubation; Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- propofol: required induction of the following agent in ICU patient
  Interventions: Procedure: induction type for intubation in ICU
- ketamine: required induction of the following agent in ICU patient
  Interventions: Procedure: induction type for intubation in ICU
- ethomidate: required induction of the following agent in ICU patient
  Interventions: Procedure: induction type for intubation in ICU
- midazolam: required induction of the following agent in ICU patient
  Interventions: Procedure: induction type for intubation in ICU

INTERVENTIONS:
Procedure: induction type for intubation in ICU — Clinical data documented throughout the course of hospitalization will be retrieved and analyzed.

SUMMARY:
The aim of this retrospective cohort study is to compare the safety and efficacy of induction agents for tracheal intubation in critically ill adult patients.

DETAILED DESCRIPTION:
Endotracheal intubation is an accepted procedure to optimize oxygenation and ventilation and reduce the risk of aspiration for critically ill patients, essential for their management and survival across various settings, including prehospital care, emergency departments (EDs), and intensive care units (ICUs). Despite advancements, peri-intubation complications and hemodynamic instability, which are associated with increased mortality rates, remain a concern. These risks are exacerbated by pathophysiological factors in critically ill patients compared to those undergoing intubation in surgical settings .

A recent international, multicentre, prospective cohort (INTUBE) study of 2964 critically ill patients undergoing tracheal intubation in the ICU, emergency department, or inpatient wards in 29 countries across five continents reported that the most frequently used agents for induction were Propofol (41.5%), Midazolam (36.4%), Etomidate (17.8%), and Ketamine (14.2%).

The choice of induction agent for intubation may have the potential to minimise or exacerbate complication and mortality. Although considerable research has been carried out, critical central question concern which induction agent is most effective in minimizing cardiovascular instability during intubation. As Kotani and Risotto declared in their recent systematic review, the available findings are insufficient to support conclusive statements. Further studies are needed to identify the optimal agent and dosage, taking into account patient variability and concurrent therapeutic interventions.

Understanding the impact of induction agent selection in critically ill patients has the potential to guide clinical practice in emergency and intensive care settings. Identifying agents with improved survival and prognosis would optimize patient management and inform decision-making for airway management in this vulnerable population. Moreover, delineating which agents exert minimal adverse effects on mortality and prognosis may provide valuable insight for anesthesiologists, intensivists, emergency medicine physicians, and trauma physicians.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to the surgical ICU for critical care
* Administration of one of the studied induction agents
* Availability of complete clinical data

Exclusion Criteria:

* Age < 18 years
* Absence of documented induction agent administration
* Incomplete or missing medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU admitted, critically ill patients The study population will include critically ill trauma patients aged 18 years and older who were admitted to the surgical intensive care unit
Sampling Method: Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome will be all-cause mortality at day 7 following tracheal intubation | day 7
  mortality at day 7

SECONDARY OUTCOMES:
Peri-intubation cardiovascular collapse | perioperatively
  occurrence after induction
Clinical course outcomes | days
  hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: TOLGA SARAÇOĞLU, Prof,MD, Principal Investigator — Florida University Jacksonville
Locations (1):
- UF Health Jacksonville (Shands Hospital), Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No